CLINICAL TRIAL: NCT06265740
Title: Early Diagnosis of Premature Births by Analysis of the Vaginal Microbiota
Acronym: PREMABIOTE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RBHP 2023 GALLOT (PREMABIOTE); 2023-A02466-39 (Other: 2023-A02466-39)
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Premature Birth; Vaginal Flora
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cohort of pregnant women at -risk of preterm delivery (Other): vaginal swab
  Interventions: Other: vaginal swab

INTERVENTIONS:
Other: vaginal swab — Any pregnant woman attending the obstetrics department of Clermont-Ferrand University Hospital who requires a vaginal swab (VS) for her clinical situation (routine care) will be offered the study. If the participant accepts, the usual swab will be doubled and performed simultaneously in a single procedure using two swabs. The first swab will be sent to the laboratory and used for diagnosis. The second swab will be used for microbiota analysis.

SUMMARY:
Objectives: to assess the relevance of the RiboTaxa algorithm coupled with neural network learning based on analysis of vaginal microbiota metagenomic sequencing data for predicting prematurity in an identified at-risk population.

Study description: Longitudinal follow-up of a cohort of pregnant women, with collection of biological samples, and a posteriori case-control comparison based on the occurrence of an event (premature birth).

DETAILED DESCRIPTION:
There is currently no reliable clinical or biological diagnosis to predict premature birth. Recent work using metagenomic data analysis coupled with artificial intelligence approaches suggests that there may be a vaginal microbiota signature during pregnancy that correlates with the occurrence of preterm birth. The aim of the study is to use biological samples to confirm the identification of these vaginal microbiota signatures as a means of predicting preterm birth.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women Admitted to the Clermont-Ferrand University Hospital maternity ward from 14 weeks' gestation onwards
* For threat of preterm birth (PTB) characterized by contractile activity and/or cervical changes, or for premature rupture of fetal membranes (PROM)
* And in need of vaginal swabbing
* Single or multiple pregnancy
* Able to understand and object to the study
* Covered by a French social security scheme.
* Give informed consent for the study

Exclusion Criteria:

* Patient under guardianship, curatorship or safeguard of justice
* Patient having received antibiotic therapy in the 2 weeks prior to admission

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03-29 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Early diagnosis of preterm birth using vaginal microbiota analysis | at birth
  prematurity yes/no (define by birth <37WG)

CONTACTS AND LOCATIONS:
Overall Officials: Denis Gallot, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France